CLINICAL TRIAL: NCT04235907
Title: Telerehabilitation Following Ankle Fractures: A Pilot Study
Brief Title: Telerehabilitation Following Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Foundation for Orthopedic Trauma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00210272
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Ankle Fractures
Keywords: Rehabilitation; Telerehabilitation
MeSH Terms: conditions — Ankle Fractures | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physical Therapy (Active Comparator): Patients will be given a prescription to see a physical therapist and a paper-based rehabilitation protocol. Patients will be allowed to receive physical therapy at a location of patients' choosing. This arm represents the current standard of care.
  Interventions: Other: Standard rehabilitation
- Telerehabilitation (Active Comparator): Patients will be given access to a website containing instructions with pictures and videos for the exercises patients are to complete as part of patients' rehabilitation. Patients will not be given a prescription to physical therapy. Patients in this group will receive weekly calls from a physical therapist during weeks 6-12 post-operatively.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Internet-guided rehabilitation with weekly phone calls from a physical therapist.
  Arms: Telerehabilitation
Other: Standard rehabilitation — Prescription for physical therapy and a printed list of exercises to complete.
  Arms: Traditional Physical Therapy

SUMMARY:
Background and Purpose: Ankle fractures represent one of the most common fractures in North America. Surgical fixation is often required in the presence of dislocation or instability and has been shown to have a high rate of success. Following surgical fixation, physical therapy is commonly utilized to assist in regaining function. Advice alone has been shown to be non-inferior to traditional physical therapy for patients post-ankle fracture in two studies. The results of these studies have yet to be repeated in the US. It is the intent of this study to investigate the feasibility of a large clinical trial comparing the results of traditional physical therapy and an internet-based telerehabilitation program. Following surgical repair of ankle fractures, patients will be randomized to traditional rehabilitation or telerehabilitation. Telerehabilitation may represent an alternative patient option to traditional physical therapy following ankle fracture repair. The results of this study will inform the design of larger multi-site clinical trials investigating the effectiveness of telerehabilitation for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Bimalleolar or trimalleolar fracture
* Repaired with open reduction internal fixation technique
* Must have access to computer, tablet, or smart phone with internet access

Exclusion Criteria:

* Severe soft tissue damage associated with injury
* Physical or mental conditions that will affect patient's ability to participate in independent rehabilitation
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in self-reported function | At 2 weeks, 6 weeks, 12 weeks, 6 months and 12 months
  Measured by the Lower Extremity Functional Scale, a patient-reported function of the lower extremity. Scores range from 0-80 with lower scores indicating increased impairment levels.

SECONDARY OUTCOMES:
Change in self-reported quality of life | At 2 weeks, 6 weeks, 12 weeks, 6 months and 12 months
  Measured using the Veterans RAND 12-Item Health Survey. This is a 12-Item global health questionnaire with a physical and mental component scores. Utilizes a t-score method standardized to the US population. Positive t-scores indicate better than average quality of life and negative t-score values represent lower than average quality of life.
Change in pain as assessed by the Brief Pain Inventory short form | At 2 weeks, 6 weeks, 12 weeks, 6 months and 12 months
  Measured using the Brief Pain Inventory short form. This is a 15-item questionnaire resulting in scores for pain severity and pain interference. Each of these is scored 0-10 with higher scores indicating increased pain severity/interference.
Patient Satisfaction as assessed by a 0-10 satisfaction scale | 6 months
  Patient reported measure of satisfaction with treatment received and progress made while recovering from injury. Will be measured on a scale of 0-10, with higher scores indicating increased satisfaction with treatment.
Out of pocket cost | 6 months
  Patient reported estimate of patients' out of pocket costs associated with rehabilitation.
Travel time (hours) | 6 months
  Patient reported estimate of time spent traveling to and from rehabilitation appointments.
Fear of pain with movement as assessed by the Tampa Kinesiophobia Scale | 2 weeks
  17-Item patient questionnaire assessing fear of movement. Scores range from 17-68 with higher scores indicating increased fear of pain with movement.
Self-Efficacy for Home Exercise Program as assessed by a 12-Item questionnaire | 2 weeks
  12-Item questionnaire assessing self-efficacy for completing assigned home exercises. Scored 0-72 with higher scores indicating increased self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin H McLaughlin, DPT, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland